CLINICAL TRIAL: NCT04932733
Title: Effects of a Single Session of Knee Isometric Exercises on Blood Pressure in Healthy Elderly: A Clinical Controlled Trial
Brief Title: Isometric Exercises in Healthy Elderly Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salameh Aldaja (Other)
Responsible Party: Sponsor-Investigator, Salameh Aldaja, Associate Professor, Isra University, Jordan
Organization: Isra University, Jordan (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 337-1/1
Record Dates: First submitted 2021-06-06; First posted 2021-06-21 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: Blood pressure; Isometric exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elderly isometric exercise (Experimental): Quadriceps isometric exercise.
  Interventions: Other: Exercises
- Young isometric exercise (Active Comparator): Quadriceps isometric exercise.
  Interventions: Other: Young isometric exercise

INTERVENTIONS:
Other: Exercises — The elderly participants in the experimental group underwent a single session of 5-minute quadriceps isometric exercise. The participant was asked to take a rest of 10 minutes before performing the exercise. After that, the exercise was performed from a long-sitting position.
  Other Names: Elderly isometric exercise
  Arms: Elderly isometric exercise
Other: Young isometric exercise — The young participants in the experimental group underwent a single session of 5-minute quadriceps isometric exercise. The participant was asked to take a rest of 10 minutes before performing the exercise. After that, the exercise was performed from a long-sitting position.
  Arms: Young isometric exercise

SUMMARY:
A total of 58 participants were selected and divided into two groups equally, namely, elderly, and young groups with the age groups of 60-80 years and 20-30 years, respectively. The Heart Rate (HR), Respiratory Rate (RR), Blood Pressure (BP), Oxygen Saturation (SaO2), and Mean Arterial Pressure (MAP) for each participant were assessed before and after the treatment session.

DETAILED DESCRIPTION:
The elderly participants in the experimental group and the young participants in the control group underwent a single session of 5-minute quadriceps isometric exercise. The participant was asked to take rest of 10 minutes before performing the exercise. After that, the exercise was performed from a long-sitting position.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were normotensive males and females in the above age groups.

Exclusion Criteria:

* Participants with a chronic history of alcohol, smoking, resting tachycardia (>100 beats per min), hypertension, history of any other cardiovascular disorders, any peripheral vascular disease, those on a regular exercise program, and uncooperative participants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure (BP) | Change from baseline blood pressure at 1 day
  Both systolic and diastolic blood pressures were measured by a trained physiotherapist in the right upper arm using an appropriate-sized cuff at the baseline and the end of the intervention using an automated Dinamap MPS Select device (Johnson & Johnson, New Brunswick, NJ).

SECONDARY OUTCOMES:
Respiratory Rate (RR) | Change from baseline respiratory rate at 1 day
  Respiratory rate was assessed by visually observe for 30 seconds and multiply observed breaths by 2 to obtain breaths per minute (BPM).
Oxygen Saturation (SaO2) | Change from baseline oxygen saturation at 1 day
  Oxygen saturation was recorded using a finger pulse oximeter. The sensor was placed on the right index finger, and the values were recorded after at least two minutes.
Heart Rate (HR) | Change from baseline heart rate at 1 day
  Heart rate was recorded using a finger pulse oximeter. The sensor was placed on the right index finger, and the values were recorded after at least two minutes.
Mean Arterial Pressure (MAP) | Change from baseline mean arterial pressure at 1 day
  Mean arterial pressure was calculated MAP as diastolic blood pressure (DBP) + 1/3 [systolic blood pressure (SBP) - DBP].

CONTACTS AND LOCATIONS:
Overall Officials: Salameh Aldaja, PhD, Principal Investigator — Isra University
Locations (1):
- Isra University, Amman, Jordan